CLINICAL TRIAL: NCT02198339
Title: A Phase II a, Double-Blind, Randomised, Group Sequential Adaptive Assignment Design Trial to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Seven Fixed Doses of Intravenous BIBN 4096 BS Ranging From 0.1 to 10.0 mg Versus Placebo in the Treatment of a Single Attach of Acute Migraine Headache
Brief Title: Efficacy, Safety, Tolerability and Pharmacokinetics of BIBN 4096 BS Versus Placebo in the Treatment of a Single Attack of Acute Migraine Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1149.2
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

ARMS (2):
- BIBN 4096 BS - ranging dose (Experimental): sequential adaptive design, allocation of verum treated patients to dose groups not fixed in advance
  IV infusion over 10 minutes
  Interventions: Drug: BIBN 4096 BS
- Placebo (Placebo Comparator): IV infusion over 10 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBN 4096 BS
  Arms: BIBN 4096 BS - ranging dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Efficacy, Safety, Tolerability and Pharmacokinetics of BIBN 4096 BS in patients with a single acute migraine attack with or without aura

ELIGIBILITY:
Inclusion Criteria:

* Man and women with an acute onset of acute migraine headache with or without aura of moderate to severe intensity
* Established diagnosis of migraine (with or without aura) according to International Headache Society (IHS) criteria for >= 1 year; age of onset <= 50 years
* Current age is 18-65 years
* Study drug treatment to begin in less than 6 hours of the onset of migraine headache which is not spontaneously improving. Time of awakening with a migraine headache is considered as time of onset provided no headache was present prior to sleep
* History of 1 to 6 migraine headaches per month for the preceding 6 months
* Ability to give written informed consent in accordance with International Committee on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation

Exclusion Criteria:

* Use of prescription and non-prescription medications for migraine prophylaxis within 2 weeks prior to treatment including Selective Serotonin Reuptake Inhibitors (SSRIs) (except fluoxetine which should have a 6 weeks washout), flunarizine (which should have a 4 week washout) and Mono-amino-oxidase-inhibitors drugs (MAOIs)
* Use of paracetamol (acetaminophen), aspirin, Non-steroidal anti-inflammatory drugs (NSAIDS), barbiturates or anti-emetics within 12 hours of taking study drug or of any 'triptan', ergotamine preparation or opiate analgesics within 48 hours prior to study drug administration or the use of analgesics > 10 days/months
* History of significant medical (i.e. coronary artery disease by history, renal failure), neurological (including epilepsy and structural brain lesions) or psychiatric disorders
* History, clinical evidence or screening or baseline electrocardiogram suggestive of cardiovascular disease including ischemic heart disease, Prinzmetal angina, coronary vasospasm, history of atherosclerotic heart disease of cardiac arrhythmia
* History of known hypertension
* History of basilar, ophthalmoplegic or hemiplegic migraine headaches or non-migraine headaches (e.g. tension-type headaches) occurring on average >= 10 days per month for the preceding 6 months
* History of treatment resistance migraine attacks defined as a lack of response to a range of commonly used acute anti-migraine compounds
* Females who are nursing or pregnant (as determined by a serum pregnancy test at screening and a urine pregnancy test at baseline) or of childbearing potential (any woman who is not at least 1 year post-menopausal or surgically sterile is considered to be of childbearing potential) and not using a medically approved method of birth control as defined by local country requirements
* Baseline systolic BP >= 160 mmHg or diastolic BP >= 100 mmHg
* Any daily intake of prescribed medication within 2 weeks prior to randomization for diseases in the investigator's judgment that would contraindicate participation in the trial
* History of Raynauds' disease
* A recent history (six months) of current evidence of alcohol or recreational drug abuse as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM- IV) (R97-1072)
* Post or present medical conditions that would keep administration of study mediation from being in the patient's best interest in the judgment of the clinical investigator
* Unwillingness or inability to comply with the protocol (e.g. the patient cannot read or write and does not have another person to assist in completing the diary; the patient cannot be followed for 1 weeks). Patients unable to give informed consent are to be excluded from participation in the trial. Patients with legally appointed custodian can not be enrolled in the trial. In case of doubt an independent psychiatrist should testify that the patient is able to give informed consent
* Use of another investigational drug within a time span of at least ten half-lives but never less than 1 month. Concurrent participation in another investigational protocol
* Prior exposure to BIBN 4096 BS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 1999-02; Primary Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Headache Response measured on a four-point scale | 2 hours post start of infusion

SECONDARY OUTCOMES:
Headache Response measured on a four-point scale | 30 min, 1, 4 and 24 hours post start of infusion
Headache Free measured on a four-point scale | 30 min, 1, 2, 4 and 24 hours post start of infusion
Maintenance of Headache Response measured on a four-point scale | up to 24 hours post start of infusion
Relief of associated symptoms | 30 min, 1, 2, 4 and 24 hours post start of infusion
Occurence of Meaningful Relief measured by stopwatch | up to 4 hours post start of infusion
Time to Meaningful Relief measured by stopwatch | up to 4 hours post start of infusion
Clinical Disability measured on four-point scale | 30 min, 1, 2, 4 and 24 hours post start of infusion
Use of rescue medication | within 24 hours post start of infusion
Time to use of rescue medication | within 24 hours post start infusion
Number of patients with adverse events | up to day 9
AUC (Area under the concentration time curve of the analyte in plasma) | up to 4 hours post start of infusion
Cmax (Maximum observed concentration of the analyte in plasma) | up to 4 hours post start of infusion
Qualified Headache Response measured on four-point scale | up to 24 hours post start of infusion
Time to sustained Headache Response | up to 24 hours post start of infusion
Worsening/Recurrence of Headache pain | 2 - 24 hours post start of infusion
Tmax (Time to maximum concentration of the analyte in plasma) | up to 4 hours post start of infusion